CLINICAL TRIAL: NCT06588972
Title: Analgesic Effects of a Treatment With Cannabis Sativa Extract in Patients With Knee Osteoarthritis - CANOA (Cannabis for Osteoarthritis)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Latin American Integration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CANOA
Record Dates: First submitted 2024-04-12; First posted 2024-09-19 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: OSTEOARTHRITIS OF THE KNEE
Keywords: Osteoarthritis; Pain; Cannabinoids; Cannabinoid safety; Tetrahydrocannabinol; Cannabidiol
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Placebo Comparator): placebo (solution of Medium Chain Triglycerides, without any active ingredient)
  Interventions: Dietary Supplement: Medium Chain Triglyceride solution
- Group 2 (Experimental): Cannabis sativa extract with a CBD (45 mg/day)
  Interventions: Other: Cannabis Sativa

INTERVENTIONS:
Dietary Supplement: Medium Chain Triglyceride solution — Placebo
  Arms: Group 1
Other: Cannabis Sativa — Group 2: Cannabis sativa extract with CBD (45mg/day).
  Arms: Group 2

SUMMARY:
Osteoarthritis (OA) is the most prevalent joint disease in humans, often causing disability in affected individuals, especially the elderly. OA is characterized by mechanical joint pain, crepitus and short-term post-immobilization stiffness. OA pain has a variable pathophysiology and, despite the many pharmacological options available, its treatment is often ineffective and has significant side effects. The search for more effective and safer treatments is therefore essential in the field of OA. Among the possible treatments are substances derived from cannabis. Cannabis plants have been used for various purposes by humankind for thousands of years. Its best-known species, Cannabis sativa, has more than a hundred substances called cannabinoids or, more specifically, phytocannabinoids, the most important of which is cannabidiol (CBD). Although many pre-clinical studies indicate the usefulness of phytocannabinoids, clinical evidence for their application is currently scarce. Therefore, this project aims to investigate the effects of a CBD-rich extract of Cannabis sativa on the pain of patients with knee OA, as well as the possible adverse events of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of knee osteoarthritis, according to the ACR classification criteria (ALTMAN, 1986);
* Have a moderate or high level of pain induced by osteoarthritis (visual analog scale scale equal to or greater than 5);
* Voluntarily agree to take part in the study by signing the Informed Consent Form (ICF);
* For women of reproductive age, a negative Beta-HCG test, and use of a contraceptive method throughout the study.
* For women of reproductive age, a negative Beta-HCG test, and use of a contraceptive method throughout the study and 3 months after its conclusion.
* Age range of thirty (30) to seventy (70) years.

Exclusion Criteria:

* People with heart failure, hypertension or any heart disease;
* People with chronic kidney disease or liver failure;
* Patients with chronic inflammatory diseases;
* Patients with severe psychiatric illnesses, such as severe mood disorders and psychotic disorders;
* Current use of cannabinoids by any route of administration.
* Pregnant women
* Lactating women

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Pain levels | 2 months
  Change in pain levels, according to the score in the "pain" domain of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), using the Likert scale to assign a value to the answers obtained from the participants. The pain levels according to the score are 0-8 mild, greater than 8-14 moderate, greater than 14- 20 high.

SECONDARY OUTCOMES:
Short Form Health Survey (SF-12) | 2 months
  Change in the Short Form Health Survey (SF-12) quality of life scores, according to the "maximal walking" and "activities of daily living" domains, where a score of 0 is the worst quality of life and 100 the best.
Depression | 2 months
  Changes in levels of depression using the Beck Depression scale. Changes in depression levels using the Beck depression scale. The disease level values range from 0-9 indicating that the individual is not depressed, 10-18 indicating mild to moderate depression, 19-29 indicating moderate to severe depression and 30-63 indicating severe depression.
Adverse events | 2 months
  presence of adverse events (AE) - proportion of patients with AE in the placebo and intervention groups;
Serious adverse events | 2 months
  presence of serious adverse events (AEs) - description of the serious AEs that may appear in each group.
Change in sleep quality | 2 months
  The Pittsburgh scale was used to see if there was any change in the participants' quality of sleep. The scale used classifies sleep quality as follows:
  * Good 0-4
  * Bad -10
  * Presence of sleep disturbance greater than 10
Renal Function Panel | 2 months
  Used as form to identify any renal impairment in pacientes that could result in any need of adjusting the dose or need to leave the study.
Visual Analogue Scale (VAS) | 2 month
  It is used in the healthcare field to measure the intensity of pain a person feels, usually on a scale from 0 to 10, where 0 means 'no pain' and 10 means 'the worst pain imaginable
Hepatic Panel | 2 month
  Used to monitor liver function in patients, as pacientes are receiving an oil-based medication that may overload the liver.

CONTACTS AND LOCATIONS:
Overall Officials: Francisney P Nascimento, 1, Study Director — Federal University of Latin American Integration
Locations (1):
- Federal University of Latin American Integration, Foz do Iguaçu, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mojoli A, Haider O, Fakih Y, Luz Goncalves MV, Zepeda Rojas B, Xaia G, Krefta E, Bicca MA, Lopes de Mari T, Ferreira CF, Cezar-Dos-Santos F, Toci AT, Nascimento FP. Effects and safety of a CBD-rich Cannabis sativa oil in knee osteoarthritis: a double-blind, randomized, placebo-controlled trial - CANOA - cannabis for osteoarthritis. Front Pharmacol. 2025 Dec 19;16:1657065. doi: 10.3389/fphar.2025.1657065. eCollection 2025. PMID 41487518